CLINICAL TRIAL: NCT02395354
Title: Comparative Prospective Multicenter Randomized Study of Endoscopic Treatment of Stenosis in Crohn´s Disease: Metal Self-expanding Prosthesis Balloon Dilatation
Brief Title: Comparative Prospective Multicenter Randomized Study of Endoscopic Treatment of Stenosis in Crohn´s Disease
Acronym: PROTDILAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grupo Espanol de Trabajo en Enfermedad de Crohn y Colitis Ulcerosa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ProtDilat-3-2013
Record Dates: First submitted 2015-03-17; First posted 2015-03-23 (Estimated); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Stenosis; Crohn's Disease; Chronic Inflammation
Keywords: Endoscopic treatment; Stenosis; Crohn's Disease; balloon dilatation; self-expanding metallic stent; chronic transmural inflammation; steady narrowing of the intestinal lumen
MeSH Terms: conditions — Constriction, Pathologic; Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placing a self-expanding metallic stent (Other): Placing a self-expanding metallic stent
  Interventions: Device: Placing a self-expanding metallic stent
- A balloon dilatation (Other): A balloon dilatation
  Interventions: Device: A balloon dilatation

INTERVENTIONS:
Device: Placing a self-expanding metallic stent — * Income on short stay unit (SSU) post-procedure
  * Light sedation by the endoscopist vs anesthetist by center
  * Fully covered self-expanding metal stents Tae Woong Medical® type; prosthesis size at the endoscopist discretion
  * Clips can be placed at the distal end of the prosthesis according to the endoscopist.
  * Prosthesis removal time in 4 weeks.
  Arms: Placing a self-expanding metallic stent
Device: A balloon dilatation — * Income on short stay unit (SSU) post-procedure
  * Light sedation by the endoscopist vs anesthetist by center.
  * Pneumatic ball type CRE Boston cientific®; balloon diameter at the endoscopist discretion
  * Up to 2 expansion will be made with a minimum interval between 15-30 days between each expansion
  * It shall be deemed failure to expansion if required> 2 expansions.
  Arms: A balloon dilatation

SUMMARY:
This study will be a multicentre randomized controlled trial to assess the efficacy between balloon dilatation and self-expanding metallic stent placement for endoscopic treatment of stenosis in Crohn´s Disease.

DETAILED DESCRIPTION:
A Prospective, randomized, multicenter clinical trial.

Duration: Beginning in mid-2013 with a minimum of three years depending on the patient inclusion rate.

The participation of at least 20 hospitals in Spain with an inclusion of about 6 patients per hospital is required.

Calculation of sample size: The calculation of sample size was performed considering that the efficacy of endoscopic treatment by endoscopic stent placement is superior to endoscopic dilatation: 75% vs 50% for balloon dilation (% of patients free of therapeutic intervention -endoscopic or surgically a year follow-up).

For all 61 patients are required for each treatment group, the total of 122 patients. This calculation is made taking into account:

* Bilateral Contrast: any two samples may be superior in terms of efficacy.
* Error type I: 0.05
* Error type II: 0.20 (statistical power 80%)
* Percentage of efficacy at one year follow-up: 75% in the prosthetic group and 50% in the balloon dilatation group
* Percentage of losses: 5%.

Schedule

1. Screening Visit
2. Sheet Inclusion
3. Expansion notebook / prosthesis placement notebook
4. Monitoring Worksheet to the 7 days. Symptomatic / complications-incidents assessment.
5. Monitoring Worksheet to the 30 days. Symptomatic / complications-incidents assessment. Includes analytical. In case of placement of prostheses include prosthetic removal sheet
6. Monitoring Worksheet to the 2 months. Symptomatic / complications-incidents assessment.
7. Monitoring Worksheet to the 3 months. Symptomatic / complications-incidents assessment.
8. Monitoring Worksheet to the 4 months. Symptomatic / complications-incidents assessment
9. Monitoring Worksheet to the 5 months. Symptomatic / complications-incidents assessment
10. Monitoring Worksheet to the 6 months. Symptomatic / complications-incidents assessment. Include analytical
11. Monitoring Worksheet to the 7 months. Symptomatic / complications-incidents assessment
12. Monitoring Worksheet to the 8 months. Symptomatic / complications-incidents assessment
13. Monitoring Worksheet to the 9 months. Symptomatic / complications-incidents assessment
14. Monitoring Worksheet to the 10 months. Symptomatic / complications-incidents assessment
15. Monitoring Worksheet to the 11 months. Symptomatic / complications-incidents assessment
16. Monitoring Worksheet to the 12 months. Symptomatic / complications-incidents assessment Include analytical.
17. Final assessment.
18. Monitoring Worksheet to the recurrence. Symptomatic / complications-incidents assessment. Include analytical

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years.
* Crohn's Disease with a predominantly fibrotic stenosis de novo and / or post- surgical confirmed by endoscopic and radiological tests, accessible by endoscopy (colonoscopy).
* Patients with stenosis already known and previously treated with stent and / or dilation with> 1 Year asymptomatic
* Symptoms of intestinal partial occlusion
* Refractory to Conventional medical treatment (no response to usual therapeutic range "accelerated step-up").
* Length of stenosis <10 cm.
* Submit a maximum of 2 stenosis.
* Patient Informed consent

Exclusion Criteria:

* No patient Informed consent.
* Stenosis complicated with abscess, fistula or important activity associated with your EC not limited to the stenosis area.
* Patients with stenosis already known and previously treated with stent and / or dilation with <1 year asymptomatic.
* Pregnancy and lactation
* Any clinical situation that prevents the performance of endoscopy
* Stenosis not accessible by endoscopy
* Asymptomatic patient
* Length of stenosis ≥ 10 cm.
* Submit> 2 stenosis.
* Severe coagulation disorders (platelets <70000; INR> 1.8)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2013-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage (%) of free patients of therapeutic intervention (dilatation, prosthesis or surgery) for symptomatic recurrence at one year follow-up | one year follow-up
  To evaluate the efficacy of endoscopic treatment (prosthesis vs dilation), determined by the percentage of free patients of a new therapeutic intervention (dilatation, prosthesis or surgery) for symptomatic recurrence at one year follow-up.
  Symptomatic recurrence assessment:
  It will be performed through an obstructive symptoms scale previously described (Attar et al, Safety and efficacy of extractible self-expandable metal stents in the treatment of Crohn's disease intestinal strictures: A prospective pilot study. Inflamm Bowel Dis. 2011 Dec 11).

SECONDARY OUTCOMES:
Percentage of free patients of therapeutic intervention (dilatation, prosthesis or surgery) for symptomatic recurrence at 6 months follow-up. | At 6 months follow-up
  To evaluate the efficacy of endoscopic treatment (prosthesis vs dilation), determined by the percentage of patients free of therapeutic intervention (dilatation, prosthesis or surgery) for symptomatic recurrence at 6 months follow-up.
  Symptomatic recurrence assessment:
  It will be performed through an obstructive symptoms scale previously described (Attar et al, Safety and efficacy of extractible self-expandable metal stents in the treatment of Crohn's disease intestinal strictures: A prospective pilot study. Inflamm Bowel Dis. 2011 Dec 11).
Rate of complications related to the procedure. | one year follow-up
  Evaluate the safety and complications of both treatments
  Immediate complications related to the procedure:
  * None
  * Inhaled into the lungs.
  * Respiratory depression O2 Sat <90%
  * Cardiorespiratory arrest
  * Arrhythmia
  * Allergic reaction
  * Pain
  * Hemorrhage: self-limiting (spontaneous hemostasis) / accurate endoscopic treatment (drooling bleeding / bleeding jet).
  * Piercing: endoscopic treatment / surgery treatment
  * Exitus
  * Others
  Late complications related to the procedure:
  * Pain
  * Hemorrhage: self-limiting (spontaneous hemostasis) / accurate endoscopic treatment (drooling bleeding / bleeding jet).
  * Piercing: endoscopic treatment / surgery treatment
  * Exitus
  * Others
The procedure total costs | one year follow-up
  Evaluate the costs of both treatments
  Study costs:
  The calculate procedure of diagnostic test (DT) cost is composed of some premises:
  * Calculate the test unit cost
  * Accounting for all costs associated with DT Direct and Indirect Costs

CONTACTS AND LOCATIONS:
Overall Officials: Carme Loras, MD, Principal Investigator — Hospital Universitari Mutua de Terrassa
Locations (1):
- Hospital Unversitari Mutua de Terrasa, Terrassa, Barcelona, Spain

REFERENCES:
- [Background] Cosnes J, Cattan S, Blain A, Beaugerie L, Carbonnel F, Parc R, Gendre JP. Long-term evolution of disease behavior of Crohn's disease. Inflamm Bowel Dis. 2002 Jul;8(4):244-50. doi: 10.1097/00054725-200207000-00002. PMID 12131607
- [Background] Rutgeerts P, Geboes K, Vantrappen G, Beyls J, Kerremans R, Hiele M. Predictability of the postoperative course of Crohn's disease. Gastroenterology. 1990 Oct;99(4):956-63. doi: 10.1016/0016-5085(90)90613-6. PMID 2394349
- [Background] Hommes DW, van Deventer SJ. Endoscopy in inflammatory bowel diseases. Gastroenterology. 2004 May;126(6):1561-73. doi: 10.1053/j.gastro.2004.03.023. PMID 15168367
- [Background] Tichansky D, Cagir B, Yoo E, Marcus SM, Fry RD. Strictureplasty for Crohn's disease: meta-analysis. Dis Colon Rectum. 2000 Jul;43(7):911-9. doi: 10.1007/BF02237350. PMID 10910235
- [Background] Hassan C, Zullo A, De Francesco V, Ierardi E, Giustini M, Pitidis A, Taggi F, Winn S, Morini S. Systematic review: Endoscopic dilatation in Crohn's disease. Aliment Pharmacol Ther. 2007 Dec;26(11-12):1457-64. doi: 10.1111/j.1365-2036.2007.03532.x. Epub 2007 Sep 28. PMID 17903236
- [Background] Thienpont C, D'Hoore A, Vermeire S, Demedts I, Bisschops R, Coremans G, Rutgeerts P, Van Assche G. Long-term outcome of endoscopic dilatation in patients with Crohn's disease is not affected by disease activity or medical therapy. Gut. 2010 Mar;59(3):320-4. doi: 10.1136/gut.2009.180182. Epub 2009 Oct 19. PMID 19840991
- [Background] Matsuhashi N, Nakajima A, Suzuki A, Yazaki Y, Takazoe M. Long-term outcome of non-surgical strictureplasty using metallic stents for intestinal strictures in Crohn's disease. Gastrointest Endosc. 2000 Mar;51(3):343-5. doi: 10.1016/s0016-5107(00)70366-x. No abstract available. PMID 10699786
- [Background] Wholey MH, Levine EA, Ferral H, Castaneda-Zuniga W. Initial clinical experience with colonic stent placement. Am J Surg. 1998 Mar;175(3):194-7. doi: 10.1016/s0002-9610(97)00285-7. PMID 9560118
- [Background] Suzuki N, Saunders BP, Thomas-Gibson S, Akle C, Marshall M, Halligan S. Colorectal stenting for malignant and benign disease: outcomes in colorectal stenting. Dis Colon Rectum. 2004 Jul;47(7):1201-7. doi: 10.1007/s10350-004-0556-5. Epub 2004 Jun 3. PMID 15164246
- [Background] Wada H, Mochizuki Y, Takazoe M, Matsuhashi N, Kitou F, Fukushima T. A case of perforation and fistula formation resulting from metallic stent for sigmoid colon stricture in Crohn's disease. Tech Coloproctol. 2005 Apr;9(1):53-6. doi: 10.1007/s10151-005-0194-5. PMID 15868501
- [Background] Bickston SJ, Foley E, Lawrence C, Rockoff T, Shaffer HA Jr, Yeaton P. Terminal ileal stricture in Crohn's disease: treatment using a metallic enteral endoprosthesis. Dis Colon Rectum. 2005 May;48(5):1081-5. doi: 10.1007/s10350-004-0865-8. PMID 15785899
- [Background] Dafnis G. Repeated coaxial colonic stenting in the palliative management of benign colonic obstruction. Eur J Gastroenterol Hepatol. 2007 Jan;19(1):83-6. doi: 10.1097/MEG.0b013e32801222f9. PMID 17206082
- [Background] Martines G, Ugenti I, Giovanni M, Memeo R, Iambrenghi OC. Anastomotic stricture in Crohn's disease: bridge to surgery using a metallic endoprosthesis. Inflamm Bowel Dis. 2008 Feb;14(2):291-2. doi: 10.1002/ibd.20268. No abstract available. PMID 17924567
- [Background] Small AJ, Young-Fadok TM, Baron TH. Expandable metal stent placement for benign colorectal obstruction: outcomes for 23 cases. Surg Endosc. 2008 Feb;22(2):454-62. doi: 10.1007/s00464-007-9453-z. PMID 17704890
- [Background] Keranen I, Lepisto A, Udd M, Halttunen J, Kylanpaa L. Outcome of patients after endoluminal stent placement for benign colorectal obstruction. Scand J Gastroenterol. 2010 Jun;45(6):725-31. doi: 10.3109/00365521003663696. PMID 20205505
- [Background] Attar A, Maunoury V, Vahedi K, Vernier-Massouille G, Vida S, Bulois P, Colombel JF, Bouhnik Y; GETAID. Safety and efficacy of extractible self-expandable metal stents in the treatment of Crohn's disease intestinal strictures: a prospective pilot study. Inflamm Bowel Dis. 2012 Oct;18(10):1849-54. doi: 10.1002/ibd.22844. Epub 2011 Dec 11. PMID 22161935
- [Background] Levine RA, Wasvary H, Kadro O. Endoprosthetic management of refractory ileocolonic anastomotic strictures after resection for Crohn's disease: report of nine-year follow-up and review of the literature. Inflamm Bowel Dis. 2012 Mar;18(3):506-12. doi: 10.1002/ibd.21739. Epub 2011 May 3. PMID 21542067
- [Background] Loras C, Perez-Roldan F, Gornals JB, Barrio J, Igea F, Gonzalez-Huix F, Gonzalez-Carro P, Perez-Miranda M, Espinos JC, Fernandez-Banares F, Esteve M. Endoscopic treatment with self-expanding metal stents for Crohn's disease strictures. Aliment Pharmacol Ther. 2012 Nov;36(9):833-9. doi: 10.1111/apt.12039. PMID 22966851
- [Derived] Loras C, Andujar X, Gornals JB, Sanchiz V, Brullet E, Sicilia B, Martin-Arranz MD, Naranjo A, Barrio J, Duenas C, Foruny JR, Busquets D, Monfort D, Pineda JR, Gonzalez-Huix F, Perez-Roldan F, Pons V, Gonzalez B, Reyes Moreno J, Sainz E, Guardiola J, Bosca-Watts MM, Fernandez-Banares F, Mayor V, Esteve M; Grupo Espanol de Trabajo de la Enfermedad de Crohn y Colitis Ulcerosa (GETECCU). Self-expandable metal stents versus endoscopic balloon dilation for the treatment of strictures in Crohn's disease (ProtDilat study): an open-label, multicentre, randomised trial. Lancet Gastroenterol Hepatol. 2022 Apr;7(4):332-341. doi: 10.1016/S2468-1253(21)00386-1. Epub 2022 Jan 20. PMID 35065738